CLINICAL TRIAL: NCT00228111
Title: Prospective Evaluation of the Additional Value of Routine Thoraco-abdominal CT in Patients That Suffered Severe Blunt Trauma of the Abdomen/Thorax
Brief Title: TRACT Study: Evaluation of the Value of Routine Thoraco-abdominal CT in Blunt Trauma Patients
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Radboud University Medical Centre
Other Study IDs: 2005/093
Record Dates: First submitted 2005-08-22; First posted 2005-09-28 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Abdominal Injuries; Thoracic Injuries
Keywords: Computed tomography; wounds and injuries,non penetrating; algorithms; Blunt trauma of the thorax and abdomen
MeSH Terms: conditions — Abdominal Injuries; Thoracic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to establish the additional effectiveness and costs of routine thoraco-abdominal computed tomography (CT) in blunt trauma patients versus conventional radiological imaging and to determine which clinical parameters predict a high additional value of routine thoraco-abdominal CT.

DETAILED DESCRIPTION:
The technological advances in computed tomography (CT), with faster image acquisition resulting in higher resolution, result in making CT a more widely and intensively used imaging modality in trauma patient care. Thoraco-abdominal CT in addition appears to have additional diagnostic value compared to conventional radiography, especially in severely injured trauma patients.

Nowadays, both clinical data and conventional radiology are used to determine which patient should undergo body CT scanning. Currently there are no widely accepted guidelines for the use of a "standard" TRAuma CT (TRACT). Although many retrospective and several prospective cohort studies have been published on this topic, the data are not sufficient to sustain evidence-based practice in decision-making.

The aim of this study is, to establish the additional effectiveness and costs of routine thoraco-abdominal CT in blunt trauma patients versus conventional radiological imaging and to determine which clinical parameters predict a high additional value of routine thoraco-abdominal CT.

Consecutive trauma patients, who are at least 16 years old and are suffering from severe injuries, undergo a standard trauma CT of the cervical spine, the thorax and abdomen after clinical evaluation and conventional radiological workup.

Clinical, conventional and computed tomographic radiological assessment, costs, therapeutic consequences and 6 months patient follow up are recorded and will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with life threatening vital problems: respiratory, circulatory (pulse > 120/min, blood pressure < 100 mmHg, refill > 4 sec, exterior blood loss > 500 ml) or neurologically (Glasgow Coma Score < 14, abnormal pupils) compromised patients.
* Patients with a revised trauma score under 12
* Patients with signs of fractures from at least two long bones
* Patients with clinical signs of flail chest/multiple rib fractures
* Patients with a clinically evident pelvic rim fracture
* Patients with signs of unstable vertebral fractures or signs of neural cord compression
* Patients involved in a high-energy injury mechanism

  * Fall from height (> 3 m)
  * As declared by prehospital emergency medical services

Exclusion Criteria:

* Patients suffering from a shock Class IIIB/IV
* Patients who need immediate neurosurgical intervention
* Pregnant patients
* Patients referred from other hospitals
* Patients who die at the emergency department

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult blunt trauma patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A.B. van Vugt, MD, PhD, Study Director — Radboud University, Dept. of Traumatology; J.G. Blickman, MD, PhD, Study Director — Radboud University, Dept. of Radiology
Locations (1):
- Radboud University, Nijmegen, Netherlands

REFERENCES:
- [Result] Brink M, Deunk J, Dekker HM, Kool DR, Edwards MJ, van Vugt AB, Blickman JG. Added value of routine chest MDCT after blunt trauma: evaluation of additional findings and impact on patient management. AJR Am J Roentgenol. 2008 Jun;190(6):1591-8. doi: 10.2214/AJR.07.3277. PMID 18492911
- [Result] Deunk J, Brink M, Dekker HM, Kool DR, van Kuijk C, Blickman JG, van Vugt AB, Edwards MJ. Routine versus selective computed tomography of the abdomen, pelvis, and lumbar spine in blunt trauma: a prospective evaluation. J Trauma. 2009 Apr;66(4):1108-17. doi: 10.1097/TA.0b013e31817e55c3. PMID 19359922
- [Result] Brink M, Deunk J, Dekker HM, Edwards MJ, Kool DR, van Vugt AB, van Kuijk C, Blickman JG. Criteria for the selective use of chest computed tomography in blunt trauma patients. Eur Radiol. 2010 Apr;20(4):818-28. doi: 10.1007/s00330-009-1608-y. Epub 2009 Sep 17. PMID 19760233
- [Derived] Brink M, de Lange F, Oostveen LJ, Dekker HM, Kool DR, Deunk J, Edwards MJ, van Kuijk C, Kamman RL, Blickman JG. Arm raising at exposure-controlled multidetector trauma CT of thoracoabdominal region: higher image quality, lower radiation dose. Radiology. 2008 Nov;249(2):661-70. doi: 10.1148/radiol.2492080169. PMID 18936319